CLINICAL TRIAL: NCT00137982
Title: Prospective Study, Randomized Controlled Trial Between Medical Treatment by Methotrexate Versus Conservative Surgical Treatment (Group 1) and Conservative Versus Radical Surgical Treatment (Group 2) to Evaluate Subsequent Fertility
Brief Title: Evaluation of Therapeutic Strategies for Treatment of Ectopic Pregnancies (EP) and Evaluation of Subsequent Fertility
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Antoine Beclere (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P030409/AOR03040
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-08

CONDITIONS: Tubal Pregnancy
Keywords: Ectopic pregnancy; Surgical treatment; Medical treatment; Fertility
MeSH Terms: conditions — Pregnancy, Tubal; Pregnancy, Ectopic

INTERVENTIONS:
Procedure: Treatment of ectopic pregnancy

SUMMARY:
Three protocols are used to treat ectopic pregnancies: medical treatment by methotrexate, conservative surgery or radical surgery. There are no data about subsequent fertility except in a cohort study. The investigators propose to evaluate the true subsequent fertility with a follow-up of 2 years, in a randomized controlled trial.

DETAILED DESCRIPTION:
The first group includes non active ectopic pregnancies defined by score or algorithm. In this case, we propose a randomized controlled trial between medical and conservative surgery. In all others clinical situations, we proposed surgery treatment. In a randomized controlled trial we compare conservative versus radical treatment. The patients are followed-up during 2 years with phone contact every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by ultra sound of ectopic pregnancy (EP)
* Patients aged > 18 years old
* Desire of future pregnancy

Exclusion Criteria:

* EP by failure of contraception
* EP associated with in vitro fertilization (IVF)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600
Dates: Start 2004-08; Study Completion 2008-07

PRIMARY OUTCOMES:
Subsequent fertility with 2 years follow-up

SECONDARY OUTCOMES:
Complications of treatments
Time of hospitalisation
Decrease curve of beta-hCG after treatment
Success rate in each group

CONTACTS AND LOCATIONS:
Overall Officials: Fernandez Hervé, PhD MD, Study Chair — Hopital Antoine Beclere
Locations (18):
- France (18):
  - Angers Hospital, Angers
  - Antoine Beclere Hospital, Clamart
  - Créteil Hospital, Créteil
  - Franco-Britannique Hospital, Levallois-Perret
  - Jeanne de Flandre Hospital, Lille
  - Hôtel Dieu, Lyon
  - Assistance Publique Hôpitaux de Marseille ; Maternité de la Conception, Marseille
  - Assistance Publique Hôpitaux de Marseille ; Hôpital Nord, Marseille
  - Maternité Régionale de Nancy, Nancy
  - Nantes Hospital, Nantes
  - Lariboisière Hospital, Paris
  - Cochin Hospital, Paris
  - Poissy Saint-Germain-en-Laye Hospital, Poissy
  - Roubaix Hospital, Roubaix
  - Charles Nicolle Hospital, Rouen
  - CMCO, Schiltigheim
  - Tours Hospital, Tours
  - Versailles Hospital ; Hôpital André Mignot, Versailles

REFERENCES:
- [Background] Fernandez H, Gervaise A. Ectopic pregnancies after infertility treatment: modern diagnosis and therapeutic strategy. Hum Reprod Update. 2004 Nov-Dec;10(6):503-13. doi: 10.1093/humupd/dmh043. Epub 2004 Sep 23. PMID 15388673
- [Derived] Bourel G, Pelletier-Fleury N, Bouyer J, Delbarre A, Fernandez H, Capmas P. Cost-effectiveness analysis of medical management versus conservative surgery for early tubal pregnancy. Hum Reprod. 2019 Feb 1;34(2):261-267. doi: 10.1093/humrep/dey352. PMID 30520964
- [Derived] Fernandez H, Capmas P, Lucot JP, Resch B, Panel P, Bouyer J; GROG. Fertility after ectopic pregnancy: the DEMETER randomized trial. Hum Reprod. 2013 May;28(5):1247-53. doi: 10.1093/humrep/det037. Epub 2013 Mar 12. PMID 23482340